CLINICAL TRIAL: NCT01836419
Title: The Clinical Efficacy of Laryngeal Mask Airway in Elderly Patients: Comparison With Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2012-0711
Record Dates: First submitted 2013-04-16; First posted 2013-04-19 (Estimated); Last update posted 2014-02-19 (Estimated); Status verified 2014-02

CONDITIONS: Minor Urologic Surgery; Lower Extremity Surgery
Keywords: classic laryngeal mask airway; elderly patients

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- young adult group (Experimental): young adult patients undergoing minor urologic surgery or lower extremity surgery
  Interventions: Procedure: classic LMA insertion
- elderly group (Active Comparator): elderly patients undergoing minor urologic surgery or lower extremity surgery
  Interventions: Procedure: classic LMA insertion

INTERVENTIONS:
Procedure: classic LMA insertion

SUMMARY:
There are some differences between elderly and young adult patients regarding the anatomy of upper airways. Elderly patients have larger upper airways than young adult patients at all pharyngeal levels as revealed by CT. Another study explained that there is a progressive descent of the larynx and epiglottis with aging, which lengthens the upper airway and possibly makes it more likely to collapse.

The aim of this study is to compare the clinical efficacy of laryngeal mask airway (LMA) in elderly patients with young adults. In this study, the investigators will measure the ease of insertion, success rate of insertion, the time of insertion, oropharyngeal leak pressure, gastric leak pressure, fiberoptic position and intraoperative complications of the classic LMA.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 20-40 and 65-85years
* ASA status 1-2
* Undergoing minor urologic surgery or lower extremity surgery
* Undergoing general anesthesia using classic LMA

Exclusion Criteria:

* Predicted difficult airway
* Increased risk of aspiration
* Gastroesophageal reflux
* Neuromuscular disease
* Significant acute or chronic lung disease

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-12; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
oropharyngeal leak pressure | 24 hours
  After successful placement of LMA, airway leak pressure was determined by adjusting the expiratory valve of the breathing circle to 40 cmH2O(fixed fresh gas flow 3 L/min) and recording the pressure when equilibrium was reached.

CONTACTS AND LOCATIONS:
Locations (1):
- Severance hospital, Seoul, Seoul, South Korea